CLINICAL TRIAL: NCT04062058
Title: A Phase II Study of Total Neoadjuvant Therapy for Locally Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jing Jin, M.D. (Unknown)
Collaborators: Beijing Hope Run (Other)
Responsible Party: Sponsor-Investigator, Jing Jin, M.D., Chinese Academy of Medical Sciences and Peking Union Medical College, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LC2018L03
Record Dates: First submitted 2019-08-18; First posted 2019-08-20 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Gastric Cancer; Neoadjuvant Therapy
Keywords: gastric cancer; neoadjuvant chemoradiotherapy; neoadjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total Neoadjuvant Chemoradiotherapy (Experimental): Total neoadjuvant chemoradiotherapy arm receives intensity-modulated neoadjuvant chemoradiotherapy (45Gy in 25 fractions) concurrently with oral S-1(40-60mg/m2, orally twice daily every weekday) followed by six cycles of SOX neoadjuvant chemotherapy and surgery
  Interventions: Radiation: SIB-IMRT; Drug: S-1; Drug: SOX; Procedure: Surgery

INTERVENTIONS:
Radiation: SIB-IMRT — 45Gy in 25 fractions using intensity-modulated radiotherapy to the radiation target
Drug: S-1 — 40-60mg/m2(according to patient's body surface area), orally twice daily every weekday concurrently with radiotherapy treatment
Drug: SOX — SOX (S-1: 40~60mg, orally twice daily on days 1 to 14, oxaliplatin 130mg/m2 intravenously on day 1, 21 days per cycle)
Procedure: Surgery — Surgery, preferred D2 lymphadenectomy

SUMMARY:
This prospective, single arm phase II study is designed to evaluate the rate of pathologic complete response of neoadjuvant chemoradiotherapy and neoadjuvant chemotherapy followed by surgery for locally advanced gastric adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven locally advanced gastric adenocarcinoma in patients staged as cT3-4N+M0
* No distant metastasis in liver,lung,bone,central nervous system(CNS),no peritoneal transplantation
* No prior abdominal or pelvic radiotherapy
* Karnofsky performance status(KPS)≥ 70, predictive life span no less than 6 months
* Patients must have normal organ and marrow function as defined below: Leukocytes: greater than or equal to 3,000 G/L; Platelets: greater than or equal to 100,000/mm3 .Hemoglobin:greater than or equal to 10g/L .Total bilirubin: within normal institutional limits; AST/ALT: less than or equal to 1.5 times the upper limit; Creatinine within normal upper limits
* Informed consent

Exclusion Criteria:

* Any prior chemotherapy or other cancer treatment prior to this protocol
* Patients with other cancer history except cervical carcinoma in situ and non-malignant melanoma skin cancer
* With any distant metastasis in liver,lung,bone,CNS,or peritoneal transplantation
* History of allergic reactions attributed to similar chemical or biologic complex to S-1 or Xeloda or Oxaliplatin
* Uncontrolled illness including, but not limited to, active infection, symptomatic heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness
* History of myocardial infarction within the past 6 months or history of ventricular arrhythmia
* History of prior radiation to the abdomen
* Pregnant or lactating females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2022-09-21 (Estimated); Study Completion 2023-09-21 (Estimated)

PRIMARY OUTCOMES:
PCR rate | 6-8 months
  Pathological response were classified into three grades.Grade I signifies that there is little shrinkage in the tumor; only mild regression in the tumor cells is observed under telemicroscope. Grade II shows gross reduction in size of the tumor and marked regression in the cancer cells microscopically, yet viable nests of cancer tissue are still visible. Grade III implies complete or almost total resolution of the tumor on exploration, and disappearance of the tumor tissue microscopically; only remnants of degenerated cancer cells can be seen (so-called ghost cancer cells).

SECONDARY OUTCOMES:
Acute chemotherapy/Chemoradiotherapy toxicities | 6-8 months
  chemotherapy toxicities are evaluated by NCI-CTC version 4.0 and radiotherapy toxicities are graded using the RTOG/EORTC Radiation Morbidity Scoring Schema.
surgery complications | 6-8 months
  During hospital stay and within the first 30 days after completion of surgery.
Tumor down-staging | 6-8 months
  Down-staging was considered as any stage reduction between clinical and pathologic stage.
R0 resection rate | 6-8 months
  The surgical procedure was total or subtotal gastrectomy with recommended D2 lymphadenectomy 4-6 weeks after total neoadjuvant therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China

REFERENCES:
- [Derived] Shi JM, Li N, Jiang LM, Yang L, Wang SL, Song YW, Liu YP, Fang H, Lu NN, Qi SN, Chen B, Li YX, Zhao DB, Tang Y, Jin J. A prospective phase II clinical trial of total neoadjuvant therapy for locally advanced gastric cancer and gastroesophageal junction adenocarcinoma. Sci Rep. 2024 Mar 29;14(1):7522. doi: 10.1038/s41598-024-58177-6. PMID 38553594
- [Derived] Shi J, Li N, Tang Y, Jiang L, Yang L, Wang S, Song Y, Liu Y, Fang H, Lu N, Qi S, Chen B, Li Z, Liu S, Wang J, Wang W, Zhu S, Yang J, Li Y, Zhao D, Jin J. Total neoadjuvant therapy for locally advanced gastric cancer and esophagogastric junction adenocarcinoma: study protocol for a prospective, multicenter, single-arm, phase II clinical trial. BMC Gastroenterol. 2022 Jul 28;22(1):359. doi: 10.1186/s12876-022-02440-5. PMID 35902798
- [Derived] Li N, Xiang X, Zhao D, Wang X, Tang Y, Chi Y, Yang L, Jiang L, Jiang J, Shi J, Liu W, Fang H, Tang Y, Chen B, Lu N, Jing H, Qi S, Wang S, Liu Y, Song Y, Li Y, Zhang L, Jin J. Preoperative versus postoperative chemo-radiotherapy for locally advanced gastric cancer: a multicenter propensity score-matched analysis. BMC Cancer. 2022 Feb 26;22(1):212. doi: 10.1186/s12885-022-09297-7. PMID 35219300